CLINICAL TRIAL: NCT03652961
Title: Rheumatoid Arthritis Memory B Cells and Abatacept (RAMBA)
Brief Title: Rheumatoid Arthritis Memory B Cells and Abatacept
Acronym: RAMBA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s18-01164; NCT03700021 (obsolete NCT alias)
Record Dates: First submitted 2018-08-23; First posted 2018-08-31 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Antirheumatic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abatacept plus DMARD (Experimental): Abatacept will be used concomitantly with standard of care disease-modifying anti-rheumatic drugs (DMARDs), other than tumor necrosis factor (TNF) antagonists or Janus kinase (JAK) inhibitors.
  Intravenous (IV) Abatacept will be administered as a 30-minute IV infusion utilizing weight range-based dosing:
  1. Less than 60 kg: 500 mg
  2. 60 to 100 kg: 750 mg
  3. More than 100 kg: 1000 mg
  Following the initial IV Abatacept administration, an IV infusion will be given at Weeks 2 and 4 after the first infusion and every 4 weeks thereafter for a total of 7 Abatacept doses.
  Abatacept will be discontinued after 6 months in all patients. Patients who have flared or failed to achieve low disease activity at 6 months will exit the trial except for one post-study visit for lab work at 9 months. In patients who have achieved low disease activity, Abatacept will be held for 6 months or until a flare results while DMARD use is continued.
  Interventions: Drug: Abatacept; Drug: DMARDs

INTERVENTIONS:
Drug: Abatacept — Abatacept for reconstitution and dilution prior to intravenous (IV) administration. Each single-use vial of Abatacept for injection provides 250-mg Abatacept, maltose (500 mg), monobasic sodium phosphate (17.2 mg), and sodium chloride (14.6 mg) for administration.
Drug: DMARDs — Patients will receive methotrexate or remain on pre-existing conventional synthetic disease-modifying anti-rheumatic drug (DMARD) if already prescribed.

SUMMARY:
Single-Open Label Study to Assess Changes in the Immune Profile in Response to Treatment with Intravenous Abatacept Adults with Rheumatoid Arthritis who are Naive to Biologic Disease-Modifying Antirheumatic Drugs

DETAILED DESCRIPTION:
The immune system of patients with Rheumatoid Arthritis (RA) is different from that of people who do not have RA. The purpose of this study is to examine participants' immune cells and proteins before initiation of study medication and after initiation of treatment with an approved therapy for RA, abatacept that will be given in combination with Methotrexate and/or anti-rheumatic drugs (DMARDS) that are approved for the treatment of RA. This study will assess whether participants have clinically responded to these medications. This assessment will also include a study of whether characteristics of participants' immune systems were changed by therapy with the study drug, abatacept.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent

  1. Subject is willing to participate in the study and has signed the informed consent.
* Target Population

  1. Men or women (not nursing or pregnant) over 18 years old who have active Rheumatoid Arthritis, defined as symptoms of Rheumatoid Arthritis prior to screening and have satisfied the American College of Rheumatology/ European League Against Rheumatism 2010 criteria for the classification of Rheumatoid Arthritis prior to signing t the informed consent.
  2. Subjects must have a Disease Activity Score 28-joint count C reactive protein (CRP) or Clinical Disease Activity Index (CDAI) assessment at screening and have at least 3 tender and at least 3 swollen joints (excluding distal interphalangeal joints) at screening and at Day 1. Patients must have at least moderate disease activity {CDAI>16); Disease Activity Score and C-reactive protein test (DAS28CRP (>4.0 )].
  3. Subjects must be naive to biologic Disease-modifying antirheumatic drugs (DMARDs)
  4. Subjects must be naive to targeted synthetic DMARDs such as tofacitinib, baricitinib, and investigational therapies for RA.
  5. Subjects receiving oral corticosteroids must be on a stable dose and at the equivalent of 10 mg prednisone daily for at least 4 weeks. Subjects may not receive an intravenous (IV), intramuscular (IM) or intra-arterial (IA) administration of a corticosteroid within 4 weeks prior to screening visit or initiation of therapy
  6. Patients with prior (including discontinued) therapy with Methotrexate and/or Hydroxychloroquine are permitted as long as they meet other inclusionary criteria.
  7. Subjects must have a DAS28CRP and Clinical Disease Activity Index (CDAI) at screening and have at least 3 tender and at least 3 swollen joints (excluding distal interphalangeal joints) at screening and at Day 1.
* Age and Reproductive Status

  1. Men and women, age's 18 years (or age of majority)
  2. Women of childbearing potential (WOCBP) must have a negative serum or urine
  3. pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within
  4. 24 hours prior to the start of study drug.
  5. Women must not be breastfeeding and must agree not to breastfeed during the study and for 100 days thereafter
  6. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug (70 days) plus 30 days (duration of ovulatory cycle) for a total of 100 days post-treatment completion.
  7. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug, plus 5 half- lives of the study drug (70 days) plus 90 days (duration of sperm turnover) for a total of 160 days post-treatment completion.
  8. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However they must still undergo pregnancy testing as described in this section. Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy.
  9. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.
  10. At a minimum, subjects must agree to use one highly effective method of contraception as listed below.
* Highly effective methods of contraception

  1. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly. WOCBP and female partners of male subjects, who are WOCBP, are expected to use one of the highly effective methods of contraception listed below. Male subjects must inform their female partners who are WOCBP of the contraceptive requirements of the protocol and are expected to adhere to using contraception with their partner.

     1. Progestogen only hormonal contraception associated with inhibition of ovulation.
     2. Hormonal methods of contraception including oral contraceptive pills containing estrogen + progesterone, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena
     3. Nonhormonal IUDs, such as ParaGard
     4. Bilateral Tubal occlusion
     5. Vasectomized partner with documented azoospermia 90 days after procedure
  2. Vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success.
  3. Intrauterine hormone-releasing system (IUS)
  4. Complete abstinence- Complete abstinence is defined as the complete avoidance of heterosexual intercourse

     1. complete abstinence is an acceptable form of contraception for all study drugs and must be used throughout the duration of the study treatment (plus 5 half-lives of the investigational drug plus 30 days).
     2. It is not necessary to use any other method of contraception when complete abstinence is elected.
     3. Subjects who choose complete abstinence must continue to have pregnancy tests
     4. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.
     5. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
* Unacceptable methods of contraception

  1. Periodic abstinence (calendar, symptothermal, post-ovulation methods)
  2. Withdrawal (coitus interruptus)
  3. Spermicide only
  4. Lactation amenorrhea method (LAM)

Exclusion Criteria:

* Target Disease Exceptions

  1. Subjects with autoimmune disease other than RA [e.g., psoriasis, systemic lupus erythematosus (SLE), vasculitis, seronegative spondyloarthritis, Inflammatory Bowel Disease, Sjogren's syndrome] or currently active fibromyalgia.
  2. Prior history of or current inflammatory joint disease other than RA (such as psoriatic arthritis, gout, reactive arthritis, Lyme disease).
* Medical History and Concurrent Diseases 1.Subjects at risk for tuberculosis (TB) defined as follows:

  1. Current clinical, radiographic or laboratory evidence of active TB. Chest x-rays (posterior anterior and lateral) obtained within the 3 months prior to obtaining written informed consent will be permitted but the images must be available and reviewed by the investigator. TB testing (IFN-gamma release assay or PPD) performed in the past month prior to Screening will be accepted; however, a copy of the report must be placed in the subject binder.
  2. A history of active TB
  3. Subjects with a positive TB screening test indicative of latent TB will not be eligible for the study unless they:
  4. Have no evidence of current TB based on chest x-ray performed And they are actively being treated for TB or the site has documentation of successful prior treatment of latent TB. Treatment regimens should be dictated by local guidelines as long as the treatment dose and duration meet or exceed local health authority guidelines. 2.Subjects with recent acute infection defined as:

  <!-- -->

  1. Any acute infection within 60 days prior to randomization that required hospitalization or treatment with parenteral antibiotics.
  2. Any acute infection within 30 days prior to randomization that required oral antimicrobial or antiviral therapy. 3. Subjects with history of chronic or recurrent bacterial infection (such as chronic pyelonephritis, osteomyelitis, and bronchiectasis etc.). 4. Subjects with any history of infection of a joint prosthesis or artificial joint.

     5. Subjects who have a history of systemic fungal infections (such as histoplasmosis, blastomycosis, or coccidiomycosis). 6. Subjects with history of recurrent herpes zoster (more than 1 episode) or disseminated (more than 1 dermatome) herpes zoster or disseminated herpes simplex, or ophthalmic zoster will be excluded. Symptoms of herpes zoster or herpes simplex must have resolved more than 60 days prior to screening. 7. Subjects with history of Human Immunodeficiency Virus (HIV) infection or who tested positive for HIV 8. Subjects with history of primary immunodeficiency

  <!-- -->

  1. Subjects who have a present malignancy or previous malignancy within the last 5 years prior to screening (except documented history of cured non-metastatic squamous or basal cell skin carcinoma or cervical carcinoma in situ). Subjects who had a screening procedure that is suspicious for malignancy, and in whom the possibility of malignancy cannot be reasonably excluded following additional clinical, laboratory or other diagnostic evaluations. 10. Current clinical findings or a history of a demyelinating disorder 11. New York Heart Association (NYHA) Class III or IV heart failure 12. Any previous or current medical conditions that are warnings against the use of TNF inhibitor agents. 13. Current clinical findings of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, psychiatric, cardiac, endocrine, neurological, or cerebral disease including severe and uncontrolled infections, such as sepsis and opportunistic infections. Concomitant medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study. 14. Subjects who have received any live vaccines within 3 months of the study drug administration or are scheduled to receive live vaccines during the study. Study subjects should not be administered a live virus vaccine for a minimum of 3 months f following the last dose of study medication. Subjects who are in close contact with others who have received a live vaccine may be enrolled at the investigator's discretion. 15. Subjects who have undergone a major surgical procedure within the 60 days prior to randomization. 16. Subjects for whom 5 or more joints cannot be assessed for tenderness or swelling (i.e. due to surgery, fusion, amputation, etc.). 17.Subjects who are prisoners, or compulsory detained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-02 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Silverman, MD, Principal Investigator — NYU Langone Health; William Rigby, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F. The epidemiology of drug treatment failure in rheumatoid arthritis. Baillieres Clin Rheumatol. 1995 Nov;9(4):619-32. doi: 10.1016/s0950-3579(05)80305-x. PMID 8591645
- [Background] Hochberg MC, Spector TD. Epidemiology of rheumatoid arthritis: update. Epidemiol Rev. 1990;12:247-52. doi: 10.1093/oxfordjournals.epirev.a036058. PMID 2286222
- [Background] Markenson JA. Worldwide trends in the socioeconomic impact and long-term prognosis of rheumatoid arthritis. Semin Arthritis Rheum. 1991 Oct;21(2 Suppl 1):4-12. doi: 10.1016/0049-0172(91)90046-3. PMID 1836280
- [Background] Spector TD. Rheumatoid arthritis. Rheum Dis Clin North Am. 1990 Aug;16(3):513-37. PMID 2217956
- [Background] Zvaifler NJ. Etiology and pathogenesis of rheumatoid arthritis. In: Arthritis and Allied Conditions. Philadelphia, PA: Lea & Febiger;1993:723-736.
- [Background] Lindqvist E, Jonsson K, Saxne T, Eberhardt K. Course of radiographic damage over 10 years in a cohort with early rheumatoid arthritis. Ann Rheum Dis. 2003 Jul;62(7):611-6. doi: 10.1136/ard.62.7.611. PMID 12810421
- [Background] Boissier MC, Semerano L, Challal S, Saidenberg-Kermanac'h N, Falgarone G. Rheumatoid arthritis: from autoimmunity to synovitis and joint destruction. J Autoimmun. 2012 Sep;39(3):222-8. doi: 10.1016/j.jaut.2012.05.021. Epub 2012 Jun 16. PMID 22704962
- [Background] Bristol-Myers Squibb Abatacept Investigator Brochure, version 18, version date 13-Nov-2014
- [Background] Schiff M. Co-stimulation Therapy in Rheumatoid Arthritis: Today and Tomorrow. Curr Treatm Opt Rheumatol. 2015;1(4):334-349. doi: 10.1007/s40674-015-0029-0. Epub 2015 Sep 29. PMID 28936386
- [Background] Emery P, Burmester GR, Bykerk VP, Combe BG, Furst DE, Barre E, Karyekar CS, Wong DA, Huizinga TW. Evaluating drug-free remission with abatacept in early rheumatoid arthritis: results from the phase 3b, multicentre, randomised, active-controlled AVERT study of 24 months, with a 12-month, double-blind treatment period. Ann Rheum Dis. 2015 Jan;74(1):19-26. doi: 10.1136/annrheumdis-2014-206106. Epub 2014 Nov 3. PMID 25367713
- [Background] Pelzek AJ, Gronwall C, Rosenthal P, Greenberg JD, McGeachy M, Moreland L, Rigby WFC, Silverman GJ. Persistence of Disease-Associated Anti-Citrullinated Protein Antibody-Expressing Memory B Cells in Rheumatoid Arthritis in Clinical Remission. Arthritis Rheumatol. 2017 Jun;69(6):1176-1186. doi: 10.1002/art.40053. Epub 2017 May 3. PMID 28118534
- [Background] Kanbe K, Chiba J, Nakamura A. Immunohistological analysis of synovium treated with abatacept in rheumatoid arthritis. Rheumatol Int. 2013 Jul;33(7):1883-7. doi: 10.1007/s00296-011-2326-8. Epub 2012 Jan 3. PMID 22212411
- [Background] Gazeau P, Alegria GC, Devauchelle-Pensec V, Jamin C, Lemerle J, Bendaoud B, Brooks WH, Saraux A, Cornec D, Renaudineau Y. Memory B Cells and Response to Abatacept in Rheumatoid Arthritis. Clin Rev Allergy Immunol. 2017 Oct;53(2):166-176. doi: 10.1007/s12016-017-8603-x. PMID 28477078
- [Background] Marasco E, Aquilani A, Cascioli S, Moneta GM, Caiello I, Farroni C, Giorda E, D'Oria V, Marafon DP, Magni-Manzoni S, Carsetti R, De Benedetti F. Switched Memory B Cells Are Increased in Oligoarticular and Polyarticular Juvenile Idiopathic Arthritis and Their Change Over Time Is Related to Response to Tumor Necrosis Factor Inhibitors. Arthritis Rheumatol. 2018 Apr;70(4):606-615. doi: 10.1002/art.40410. Epub 2018 Mar 25. PMID 29316374
- [Background] Westhovens R, Robles M, Ximenes AC, Nayiager S, Wollenhaupt J, Durez P, Gomez-Reino J, Grassi W, Haraoui B, Shergy W, Park SH, Genant H, Peterfy C, Becker JC, Covucci A, Helfrick R, Bathon J. Clinical efficacy and safety of abatacept in methotrexate-naive patients with early rheumatoid arthritis and poor prognostic factors. Ann Rheum Dis. 2009 Dec;68(12):1870-7. doi: 10.1136/ard.2008.101121. Epub 2009 Jan 5. PMID 19124524

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept Plus DMARD: Abatacept will be used concomitantly with standard of care disease-modifying anti-rheumatic drugs (DMARDs), other than tumor necrosis factor (TNF) antagonists or Janus kinase (JAK) inhibitors.
  Intravenous (IV) Abatacept will be administered as a 30-minute IV infusion utilizing weight range-based dosing:
  1. Less than 60 kg: 500 mg
  2. 60 to 100 kg: 750 mg
  3. More than 100 kg: 1000 mg
  Following the initial IV Abatacept administration, an IV infusion will be given at Weeks 2 and 4 after the first infusion and every 4 weeks thereafter for a total of 7 Abatacept doses.
  Abatacept will be discontinued after 6 months in all patients. Patients who have flared or failed to achieve low disease activity at 6 months will exit the trial except for one post-study visit for lab work at 9 months. In patients who have achieved low disease activity, Abatacept will be held for 6 months or until a flare results while DMARD use is continued.
  Abatacept: Abatacept for reconstitution and dilution prior to intravenous (IV) administration. Each single-use vial of Abatacept for injection provides 250-mg Abatacept, maltose (500 mg), monobasic sodium phosphate (17.2 mg), and sodium chloride (14.6 mg) for administration.
  DMARDs: Patients will receive methotrexate or remain on pre-existing conventional synthetic disease-modifying anti-rheumatic drug (DMARD) if already prescribed.
Period: Overall Study
Arm/Group | Abatacept Plus DMARD
Started | 25
Completed | 21
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abatacept Plus DMARD
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 56.7 [25 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: CDAI Score
Description: Clinical Disease Activity Index (CDAI) is a composite index used to assess rheumatoid arthritis (RA) disease activity.
  The CDAI score is the sum of the Swollen 28-Joint Count (SJC28) + Tender 28-Joint Count (TJC) + Patient Global disease Activity (PGA, patient's assessment of overall RA disease activity on a scale 1-10 where 10 is maximal activity) + Evaluator's Global disease Activity (EGA, evaluator's assessment of overall RA disease activity on a scale 1-10 where 10 is maximal activity). The total score range is 2-76; higher scores (CDAI > 22) indicate HIgh Disease Activity.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept Plus DMARD
Number analyzed (Participants) | 21
score on a scale | 36.06 (14.59)

2. Primary Outcome: CDAI Score
Description: as for outcome 1
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept Plus DMARD
Number analyzed (Participants) | 18
score on a scale | 6.86 (5.87)

3. Primary Outcome: DAS-28 CRP Score
Description: Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) is a composite index used to assess rheumatoid arthritis (RA) disease activity.
  The DAS-28 CRP score is calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (scored on 11-point Likert scale from 0 [no disease activity] to 10 [maximum disease activity]), and high-sensitivity C-reactive protein levels (in mg/L). DAS28-CRP Scores range from 0 to 10; higher scores indicate more active disease.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept Plus DMARD
Number analyzed (Participants) | 21
score on a scale | 3.60 (1.45)

4. Primary Outcome: DAS-28 CRP Score
Description: as for outcome 3
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept Plus DMARD
Number analyzed (Participants) | 18
score on a scale | 2.61 (0.98)

5. Secondary Outcome: DAS-28 CRP Score After Abatacept Hold
Description: as for outcome 3
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept Plus DMARD
Number analyzed (Participants) | 18
score on a scale | 3.14 (2.02)

6. Secondary Outcome: CDAI Score After Abatacept Hold
Description: as for outcome 1
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept Plus DMARD
Number analyzed (Participants) | 18
score on a scale | 16.83 (18.84)

ADVERSE EVENTS:
Time Frame: 9 months
Description: Standard questionnaire at every visit
Arm/Group | Abatacept Plus DMARD
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 10/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept Plus DMARD (N=21)
URI (Respiratory, thoracic and mediastinal disorders) | 8 (10)
transient dyspnea-self resolving without treatment (Respiratory, thoracic and mediastinal disorders) | 1
Self-limited rash - transient (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT03652961/Prot_SAP_000.pdf